CLINICAL TRIAL: NCT02811536
Title: Investigation of Vascular Pathology in Eye Diseases Using Using Optical Coherence Tomography Angiography (OCT-A)
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: OCTA Bern
Record Dates: First submitted 2016-06-20; First posted 2016-06-23 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Diabetic retinopathy: Patients with various degrees of diabetic retinopathy
  Interventions: Device: optical coherence tomography angiography
- Retinal detachment: Patients with a history of retinal detachment
  Interventions: Device: optical coherence tomography angiography
- Retinal vein occlusion: Patients with a history of retinal vein occlusion
  Interventions: Device: optical coherence tomography angiography
- Arterial hypertension: Patients with a history of arterial hypertension
  Interventions: Device: optical coherence tomography angiography
- Carotid artery occlusion: Patients with a history of carotid artery occlusion
  Interventions: Device: optical coherence tomography angiography
- Age related macular degeneration: Patients with a history of Age related macular degeneration
  Interventions: Device: optical coherence tomography angiography
- Macroaneurysms: Patients with a history of retinal macroaneurysms
  Interventions: Device: optical coherence tomography angiography
- Central serous chorioretinopathy: Patients with a history of central serous chorioretinopathy
  Interventions: Device: optical coherence tomography angiography

INTERVENTIONS:
Device: optical coherence tomography angiography — Imaging with optical coherence tomography angiography

SUMMARY:
Comparison of OCTA to conventional imaging modalities for the diagnosis of eye diseases

DETAILED DESCRIPTION:
Optical coherence tomography angiography (OCTA) is a new non-invasive imaging technique that employs motion contrast imaging to high-resolution volumetric blood flow information. OCTA compares the decorrelation signal between sequential OCT b-scans taken at precisely the same cross-section in order to construct a map of blood flow. At present, level 1 evidence of the technology's clinical applications doesn't exist. The investigators plan to compare OCTA as an imaging modality to conventional imaging modalities used in clinical routine.

ELIGIBILITY:
Inclusion criteria:

Patients from the Department of Ophthalmology, University Hospital Bern requiring conventional imaging for eye disease and willing to sign informed consent Patients of 18 years or older

Exclusion criteria:

Patients not willing or able to sign informed consent Patients younger than 18 years Patients with epilepsy Patients having had photodynamic therapy within the last 48 hours prior to imaging with OCTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with a history of clinically diagnosed retinal diseases, including but not limited to age-related macular degeneration, diabetic retinopathy, retinal vein occlusion, macular macroaneurysma, and diabetic macular edema and healthy individuals undergoing ophthalmic Imaging in Routine clinical practice will be included
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of the sensitivity and specificity of OCTA | 2 years
  The primary objective of this observational study is to evaluate the sensitivity and specificity to diagnose vascular abnormalities with OCTA compared to conventional imaging methods. The main parameter that will be assessed is area of nonperfusion of the retina. The incidence (binary) of nonperfusion areas will be assessed in OCTA and compared to conventional imaging methods such as fluorescein angiography.

SECONDARY OUTCOMES:
Evaluation of the intra-and inter-reader reproducibility of the diagnosis of vascular abnormalities using OCTA | 2 years
  The primary objective of this observational study is to evaluate the sensitivity and specificity to diagnose vascular abnormalities with OCTA compared to conventional imaging methods. The main parameter that will be assessed is area of nonperfusion of the retina. The incidence (binary) of nonperfusion areas will be assessed in OCTA and compared to conventional imaging methods such as fluorescein angiography.
OCTA and Fundus color photographs | 2 years
  Evaluation whether pathological changes seen in OCT or color fundus photography correlate with changes seen in OCTA
Subgroup analysis | 2 years
  Subgroup analysis will be performed with patients suffering from diabetic retinopathy, artery occlusion, carotid stenosis, retinal detachment, vein occlusion, age related macular degeneration, retinal changes from arterial hypertension, retinal macroaneurysms and uveitis.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zinkernagel, Prof.MD PhD, Study Chair — Inselspital, University Clinic for Ophthalmology
Locations (1):
- Inselspital Bern, Department of Ophthalmology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian M, Zeng G, Zinkernagel M, Tappeiner C, Wolf S, Munk MR. Assessment of choriocapillaris and choroidal vascular changes in posterior uveitis using swept-source wide-field optical coherence tomography angiography. Br J Ophthalmol. 2024 Feb 21;108(3):386-390. doi: 10.1136/bjo-2022-322209. PMID 36627172
- [Derived] Tian M, Tappeiner C, Zinkernagel MS, Huf W, Wolf S, Munk MR. Evaluation of vascular changes in intermediate uveitis and retinal vasculitis using swept-source wide-field optical coherence tomography angiography. Br J Ophthalmol. 2019 Sep;103(9):1289-1295. doi: 10.1136/bjophthalmol-2018-313078. Epub 2018 Dec 11. PMID 30538102